CLINICAL TRIAL: NCT04412252
Title: A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY ASSESSING THE SAFETY AND EFFICACY OF TOFACITINIB IN HOSPITALIZED PARTICIPANTS WITH COVID-19 PNEUMONIA WHO ARE RECEIVING STANDARD OF CARE THERAPY
Brief Title: Safety and Efficacy of Tofacitinib in Hospitalized Participants With COVID-19 Pneumonia Who Are Receiving Standard of Care Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the pursuit of other SARS-CoV-2-related research including alternative trials with tofacitinib, this trial was canceled prior to subject enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921377
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: COVID-19; Pneumonia; SARS-CoV-2; Novel Coronavirus
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tofacitinib (Experimental): Participants will receive tofacitinib 10 mg twice per day for 14 days and standard of care therapy.
  Interventions: Drug: Tofacitinib
- Placebo (Placebo Comparator): Participants will receive tofacitinib-matching placebo twice per day for 14 days and standard of care therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tofacitinib — 10 mg tofacitinib administered as two 5 mg tablets or solution taken orally twice daily for 14 days
  Other Names: xeljanz
  Arms: Tofacitinib
Other: Placebo — Tofacitinib-matching placebo administered as tablets or solution taken orally twice daily for 14 days
  Arms: Placebo

SUMMARY:
The study is designed as a multicenter, randomized, double-blind, placebo-controlled, parallel group study of the safety and efficacy of tofacitinib in hospitalized adult participants with COVID-19 pneumonia who are receiving SoC therapy and who are not on HFNC, noninvasive ventilation, invasive mechanical ventilation, or ECMO on Day 1 at the time of randomization.

Participants with laboratory confirmed SARS-CoV-2 infection as determined by a positive PCR or other commercially available or public health assay, who have agreed to participate will be screened within 48 hours after hospitalization to determine eligibility. This should be completed within 48 hours prior to Day 1.

Eligible participants will be randomized on Day 1 in a 1:1 ratio to the tofacitinib treatment group or the placebo treatment group and will receive treatment for up to 14 days, or until discharge from the hospital, whichever is earlier. If a participant requires intubation prior to the end of the 14-day treatment period, they will continue to receive tofacitinib or matching placebo until Day 14 (or until discharge from the hospital, if earlier than Day 14), if clinically appropriate.

Participants will be assessed daily (up to Day 28) while hospitalized for clinical, safety, and laboratory parameters. Follow-up visits will occur on Day 28, 28 to 35 days after the ET/ED/EOT visit, and on Day 60.

An independent, external DSMB will be convened to oversee the safety of participants and make recommendations regarding the conduct of the trial in accordance with the Charter.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years. A female is eligible if she is not pregnant or breastfeeding. WOCBP must use 2 highly effective forms of contraception.
* Participants with laboratory-confirmed novel coronavirus (SARS-CoV-2) infection prior to Day 1.
* Participants with evidence of COVID-19 pneumonia assessed by radiographic imaging (chest x ray or chest CT scan).

Exclusion Criteria:

* Require HFNC, non-invasive ventilation, invasive mechanical ventilation, or ECMO on Day 1 at the time of randomization.
* Have history of or current thrombosis. Only if current thrombosis is suspected, imaging testing is recommended (e.g. CTPA or per local guidance) to exclude thrombosis.
* Have a personal or first degree family history of blood clotting disorders.
* Participants who are immunocompromised, with known immunodeficiencies, or taking potent immunosuppressive agents (e.g. azathioprine, cyclosporine).
* Participants with any current malignancy or lymphoproliferative disorders that requires active treatment.
* Suspected or known active systemic bacterial, fungal, or viral infections (with the exception of COVID-19).
* Severe hepatic impairment, defined as Child-Pugh class C.
* Severe anemia (hemoglobin < 8 g/dL)
* ANY of the following abnormalities in clinical lab tests at screening, confirmed by a single repeat, if deemed necessary: ALC < 500 cells/mm3, ANC < 1000 cells/mm3
* Known allergy to tofacitinib

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-06 (Estimated); Primary Completion 2020-09-16 (Estimated); Study Completion 2020-10-18 (Estimated)

PRIMARY OUTCOMES:
Clinical status using ordinal scale | Day 28
  Death or respiratory failure (1, 2, or 3, on an 8-point ordinal scale of disease severity) at Day 28. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.

SECONDARY OUTCOMES:
Clinical status using ordinal scale | Day 14
  Ordinal scale of disease severity. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Status of alive and not using mechanical ventilation or extracorporeal membrane oxygenation (ECMO) | Day 14 and Day 28
  Category 3 to 8 on an ordinal scale of disease severity. The scale is as follows: 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Status of discharged or not requiring supplemental oxygen | Day 28
  Category 5 to 8 on an ordinal scale of disease severity. The scale is as follows: 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Mortality | Day 60
  Category 1 on an ordinal scale of disease severity. The scale is as follows: 1) Death.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Hartford Hospital (HH), Hartford, Connecticut
  - University of Iowa Hospitals & Clinics Investigational Drug Services, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa
  - LSUHSC-Shreveport, Shreveport, Louisiana
  - Ochsner LSU Health Shreveport Academic Medical Center, Shreveport, Louisiana
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921377